CLINICAL TRIAL: NCT04204837
Title: Phase II Study of Nivolumab (Group 1) and Nivolumab Plus Relatlimab (Group 2) in Patients With Locally Advanced/ Metastatic Squamous Cell Carcinoma of the Skin
Brief Title: Nivolumab for Treatment of Squamous Cell Carcinoma of the Skin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Martin Laimer, MD, MSc, a.o. Univ.-Prof. Dr. med. univ., MSc, Salzburger Landeskliniken
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-587
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Squamous Cell Carcinoma of the Skin
Keywords: Nivolumab; Relatlimab
MeSH Terms: interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab (Experimental): Nivolumab will be given on Day 1 of every 14-day cycle (Q2W) at a dose of 240 mg as an IV infusion until progression, unacceptable toxicity or discontinuation for other reasons for up to 2 years.
  Interventions: Drug: Nivolumab
- Nivolumab plus Relatlimab (Experimental): Patients wil receive a fixed-dose combination of nivolumab 480 mg and relatlimab 160 mg by intravenous infusion every four weeks (Q4W) (Group 2) for up to two years after initial dosing or until PD - or absence of investigator-assessed clinical benefit
  Interventions: Drug: Nivolumab plus Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given on Day 1 of every 14-day cycle (Q2W) at a dose of 240 mg as an IV infusion until progression, unacceptable toxicity or discontinuation for other reasons for up to 2 years.
  Arms: Nivolumab
Drug: Nivolumab plus Relatlimab — Patients wil receive a fixed-dose combination of nivolumab 480 mg and relatlimab 160 mg by intravenous infusion every four weeks (Q4W) (Group 2) for up to two years after initial dosing or until PD - or absence of investigator-assessed clinical benefit
  Arms: Nivolumab plus Relatlimab

SUMMARY:
To determine the Objective Response Rate (ORR) of immunotherapy with Nivolumab (Group 1) and Nivolumab plus Relatlimab (Group 2) in patients with locally advanced/metastatic squamous cell carcinoma of the skin using Response Criteria in Solid Tumors Version 1.1 (RECIST1.1) per site assessment (Time Frame Group 2: From first dose up to 5 years)

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 years of age and older on day of signing written informed consent
2. Histologically or cytologically documented locally-advanced and/or metastatic squamous cell carcinoma of the skin (stage III/IV AJCC 2010) that is incurable
3. Archival tumor tissue available for evaluation of PD-L1 and LAG-3 expression
4. Measurable disease based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
5. Life expectancy of at least 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2
7. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to registration:

   * WBC ≥ 2000/μl
   * Neutrophils ≥ 1500/μL
   * Platelets ≥ 100 x103/μL
   * Hemoglobin > 9.0 g/dL
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

   Female CrCl = (140 - age in years) x weight in kg x 0.85/72 x serum creatinine in mg/dL Male CrCl = (140- age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL
   * AST/ALT ≤ 3 x ULN
   * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
   * Negative pregnancy test and effective contraception (Pearl-Index <1) for for women of childbearing potential (WOCBP) if the risk of conception exists
8. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration
9. Prior systemic antibiotic treatment must have been completed at least 30 days prior to stool sample collection

Exclusion Criteria:

1. Patient is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
2. Prior therapy with CTLA-4, PD-1 or LAG-3 antibodies
3. History of myocarditis, regardless of etiology
4. Troponin T (TnT) or I (TnI) > 2× institutional upper limit of normal (ULN). Participants with TnT or TnI levels between > 1× to 2× ULN will be permitted if repeat levels within 24 hours are ≤ 1× ULN. If TnT or TnI levels are between > 1× to 2× ULN within 24 hours, the participant may undergo a cardiac evaluation and be considered for treatment, based on a favorable benefit/risk assessment by the Investigator. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2× ULN, the participant may undergo a cardiac evaluation and be considered for treatment, based on a favorable benefit/risk assessment by the Investigator
5. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
6. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
7. Known additional malignancy that is progressing or requires active treatment. Patients with chronic lymphocytic leukemia that is stable under active therapy are eligible for inclusion.
8. An active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
9. Patients with serious intercurrent illness, requiring hospitalization
10. Other serious illnesses, e.g. serious infections requiring antibiotics
11. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
12. Pregnancy (absence to be confirmed by ß-HCG urinary test, minimum sensitivity 25 IU/L or equivalent units of HCG)) or lactation period
13. Women of childbearing potential (WOCBP): Refusal or inability to use effective means of contraception (Pearl-Index <1)
14. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
15. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
17. Known hypersensitivity reaction to any of the components of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 5 years
  using Response Criteria in Solid Tumors Version 1.1 (RECIST1.1) per site assessment

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 5 years
  Disease Control Rate (DCR) using Response Criteria in Solid Tumors version 1.1 (RECIST1.1) per site assessment
Duration of Response (DOR) in patients who achieve partial response (PR) or better | up to 5 years
Progression Free Survival (PFS) | up to 5 years
Overall Survival (OS) | up to 5 years
ORR and DCR for patients with PD-L1-positive tumor expression and/or positive LAG-3 expression of tumor-infiltrating cells | up to 5 years
Number and severity of adverse events | up to 5 years
DOR, PFS and OS for patients with PD-L1-positive tumor expression and/or positive LAG-3 expression of tumor-infiltrating cells | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Laimer, MD, Principal Investigator — Salzburger Landeskliniken
Locations (7):
- Austria (7):
  - Universitätsklinikum Graz - LKH, Klinische Abteilung für Onkologie, Graz
  - LKH Innsbruck Universitätsklinik für Dermatologie und Venerologie, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Universitätsklinik für Dermatologie und Allergologie der Paracelsus medizinischen Privatuniversität Salzburg, Salzburg
  - Abteilung für Haut- und Geschlechtskrankheiten, Universitätsklinikum St. Pölten Karl Landsteiner Privatuniversität für Gesundheitswissenschaften, Sankt Pölten
  - Med Uni Wien, Univ. Klinik für Dermatologie, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels